CLINICAL TRIAL: NCT04315246
Title: A Phase I/II Trial of Intracerebroventricular 177Lu DTPA Omburtamab Radioimmunotherapy for Leptomeningeal Metastasis From Solid Tumors
Brief Title: 177Lu-DTPA-Omburtamab Radioimmunotherapy for Leptomeningeal Metastasis From Solid Tumors (Breast, NSCLC, Malignant Melanoma)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business priorities
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 302
Record Dates: First submitted 2020-03-12; First posted 2020-03-19 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Leptomeningeal Metastasis; Solid Tumor, Adult
MeSH Terms: conditions — Meningeal Carcinomatosis

STUDY DESIGN:
Intervention Model Description: Patients will receive up to five cycles of intracerebroventricular 177Lu-DTPA-omburtamab. Safety and efficacy will be investigated during treatment and follow-up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 177Lu-DTPA-omburtamab (Experimental): Intracerebroventricular administration of 177Lu-DTPA-omburtamab for up to five cycles.
  Interventions: Biological: radiolabeled DPTA-omburtamab

INTERVENTIONS:
Biological: radiolabeled DPTA-omburtamab — Biological, radiolabeled DPTA-omburtamab
  Other Names: Drug: 177Lu-DTPA-omburtamab

SUMMARY:
Adults with leptomeningeal metastasis from solid tumors will be treated with 177Lu-DTPA-omburtamab, which is a radioactive labelling of a murine monoclonal antibody targeting B7-H3.

DETAILED DESCRIPTION:
Part 1 is a dose-escalation phase with a 3+3 sequential-group design in which patients will receive a dosimetry dose followed by maximum of five 5-week cycles of treatment doses of intracerebroventricular 177Lu-DTPA-omburtamab.

Part 2 is a cohort-expansion phase in which patients will receive a treatment at the recommended dose determined in Part 1, until confirmed LM progression, unacceptable toxicity, or for maximum of 5 cycles, whichever comes first; however, the total number of cycles will be determined based upon data from Part 1 (e.g., the dosimetry data) to minimize the risk of radiation necrosis and decreased neurological function End of treatment will take place within 5 weeks after the last cycle and thereafter the patients will be enter the follow-up period. The patients will be followed for up until one year after first dose (Part 1) and 2 years after first dose (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Primary ductal or lobular breast cancer, non-small cell lung cancer, or malignant melanoma
* Type I or Type II LM with a "confirmed" or "probable" diagnosis according to EANO-ESMO guidelines 2017
* Life expectancy more than 2 months, as judged by the Investigator
* ECOG Performance status 0, 1, or 2
* Acceptable hematological status and liver and kidney function
* Written informed consent obtained in accordance with local regulations
* Presence of an intracerebroventricular access device before first dosing

Exclusion Criteria:

* Obstructive or symptomatic communicating hydrocephalus
* Progressive systemic (extra-leptomeningeal) disease
* Uncontrolled life-threatening infection
* Ventriculo-peritoneal shunts without programmable valves. Ventriculo-atrial or ventriculo-pleural shunts
* Received craniospinal irradiation (for intraparenchymal or dural metastases) or intrathecal cytotoxic anti-cancer therapy less than 3 weeks prior to first dose of 177Lu-DTPA-omburtamab
* Severe non-hematologic organ toxicity; specifically, any renal, cardiac, hepatic, pulmonary, or gastrointestinal system toxicity Grade 3 or above prior to enrolment
* Grade 4 nervous system disorder. Hearing loss or stable neurological deficits due to brain tumor are allowed
* Unacceptable coagulation function prior to first dosing defined as INR Grade 2 or above
* Female of childbearing potential, who are pregnant, breast-feeding, intend to become pregnant, or are not using highly effective contraceptive methods or male who is not using highly effective contraceptive method
* Other significant disease or condition that in the investigator's opinion would exclude the patient from the trial.
* Smallest diameter of treated or untreated nodular or linear leptomeningeal metastasis >0.5 cm on MRI (Part 2 only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 1 year
  Safety will be evaluated by the incidence of AEs and SAEs graded according to CTCAE version 5.0. The maximum tolerated dose and the recommended phase 2 dose (RP2D) will be determined in Part 1
Incidence of AEs and SAEs | 2 years
  In Part 2, safety will be evaluated by the incidence of AEs and SAEs graded according to CTCAE version 5.0, at the RP2D defined in Part 1

SECONDARY OUTCOMES:
Maximum radioactivity count of lutetium-177 in blood | 2 weeks
  The time for maximum absorbed radiation dose
Elimination half-life of lutetium-177 radioactivity in blood | 2 weeks
  The time for eliminating half of the radioactivity in blood
Absorbed radiation dose of lutetium-177 in blood and cerebrospinal fluid (CSF) | 2 weeks
  Time-activity curves of radioactivity measurements in blood and CSF will be modeled to deliver absorbed doses in blood and CSF
Dosimetry analysis of lutetium-177 | 2 weeks
  Whole-body dosimetry by gamma camera scans and single-photon emission computed tomography (SPECT)
Maximum Plasma Concentration [Cmax] in CSF | 7 weeks
  Concentration of 177Lu-DTPA-omburtamab in CSF
Maximum Plasma Concentration [Cmax] in serum | 7 weeks
  Concentration of 177Lu-DTPA-omburtamab in serum
Elimination Half Life in CSF | 7 weeks
  Concentration of 177Lu-DTPA-omburtamab in CSF
Elimination Half Life in serum | 7 weeks
  Concentration of 177Lu-DTPA-omburtamab in serum
Response | 2 years
  Objective response rate (ORR) will be defined as the proportion of all evaluable patients achieving a response as the best overall response at the time of assessment
Investigator-assessed Duration of Response (DoR) | 2 years
  DoR is defined as the time from first response to LM progression
Progression-free Survival (PFS) | 2 years
  PFS is defined as the time from first treatment to date of LM progression or death from any cause, whichever comes first
Overall Survival (OS) | 2 years
  OS is defined as the time from first treatment to date of death

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Johns Hopkins, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - M.D. Anderson Cancer Center, Houston, Texas
  - The University of Washington, Seattle, Washington
- United Kingdom (2):
  - The Christie Hospital NHS Foundation Trust, Manchester
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Undecided